CLINICAL TRIAL: NCT02123160
Title: Dyadic Therapy for Mothers and Children
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of staff
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Sackler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6687
Record Dates: First submitted 2014-03-31; First posted 2014-04-25 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Depression; Behavioral Problems
Keywords: Depression; Dyadic therapy; Behavioral Problems; Child parent therapy; Affect regulation; Immune markers; Cortisol
MeSH Terms: conditions — Depression; Problem Behavior

STUDY DESIGN:
Intervention Model Description: Psychotherapy-behavioral intervention
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child Parent Psychotherapy (CPP) (Experimental): Following Time 1 (pre-treatment) assessment, mother-child patient dyads will be randomly assigned to either Child Parent Psychotherapy (CPP) treatment or control (usual treatment) group. CPP treatment will be conducted by a CPP study clinician over approximately six months (24 weekly sessions). CPP includes developmental guidance and fostering affect regulation , continuity in daily living, reciprocity between mother and child, and helping the mother and child understand themselves and each other in the context of the maternal psychiatric functioning and/or familial exposure to trauma.
  Interventions: Behavioral: Child Parent Psychotherapy (CPP)
- Usual Treatment (Active Comparator): Following Time 1 (pre-treatment) assessment, mother-child patient dyads randomized to the control group will be referred for usual treatment via referral to therapists in the community and at Columbia University Medical Center, for psychoeducation, counseling/ therapy for maternal depressive symptoms, and child behavioral/ emotional difficulties. Additionally, control patient dyads will be monitored through regular contact with the study research assistant. If the research assistant detects worsening of depressive symptoms or the presentation of new symptoms, a licensed study clinician will follow up to assess mother/ child's psychiatric functioning and make necessary referrals to alternative treatments or arrange an emergency evaluation, if needed.
  Interventions: Behavioral: Control (usual treatment)

INTERVENTIONS:
Behavioral: Child Parent Psychotherapy (CPP) — Child Parent Psychotherapy (CPP) is a multi-theoretical approach to enhance the caregiver-child relationship in the context of the caregiver's psychiatric history (e.g., depression) and/or caregiver/child exposure to traumatic events. Mother and child's in-session interactions are used to provide developmental guidance, and reinforce reciprocity between parent and child, affect regulation , continuity in daily living, and helping mother and child understand themselves and each other in the context of the maternal psychiatric functioning and/or familial exposure to trauma. When there is a history of trauma exposure for mother and/or child, mother and child create a joint narrative of the trauma, identify and address traumatic triggers, and focus on safety issues.
  Arms: Child Parent Psychotherapy (CPP)
Behavioral: Control (usual treatment) — Following Time 1 (pre-treatment) assessment, mother-child patient dyads randomized to the control group will be referred to usual treatment in the community for psychoeducation, counseling/ therapy for maternal depressive symptoms, and child behavioral/ emotional difficulties. Control patient dyads will be closely monitored through regular contact with the study research assistant and follow up by a licensed study clinician to assess mother/ child's psychiatric functioning and make necessary referrals to alternative treatments or arrange an emergency evaluation, if needed.
  Arms: Usual Treatment

SUMMARY:
This study compares the effectiveness of Child Parent Psychotherapy to that of usual care (defined as: referral to therapists in the community or Columbia University Medical Center) in improving maternal depressive symptoms and child emotional and behavioral disturbances. The investigators will recruit mothers who report being mildly to moderately depressed and their preschoolers (ages 3-5 years) who they are concerned are exhibiting emotional and/or behavioral problems.

DETAILED DESCRIPTION:
Child Parent Psychotherapy (CPP) has been demonstrated to be effective in improving mother-child attachment relationship, maternal (depression, posttraumatic stress symptoms, global symptoms of distress) and child (behavior problems, posttraumatic stress symptoms and diagnosis, cognitive and representational models) outcomes, in the context of risk factors such as maternal depression and exposure to traumatic events. It is the only treatment for preschool aged children and caregivers that seeks to affect changes at both behavioral and schematic/ cognitive levels. The investigators aim to assess the feasibility and acceptability of providing CPP as a dyadic preventive intervention for children who are displaying signs of emotional and behavioral difficulties in the context of maternal depression.

Investigators will compare the effectiveness of CPP to that of usual care (usual care defined as: referral to therapists in the community and within Columbia University Medical Center for psychoeducation, counseling/ therapy for maternal depressive symptoms, and child behavioral/ emotional difficulties) in improving maternal depressive symptoms and child emotional and behavioral problems. The investigators will recruit mothers who report being mildly to moderately depressed and their preschoolers (aged 3-5 years) who they are concerned are exhibiting emotional and/or behavioral problems.

Mother-child patient dyads will be screened via telephone to assess study eligibility. If eligible mothers and their children will complete an in-person pre-treatment assessment. After the Time 1 (pre-treatment) assessment, mother-child patient dyads will be randomly assigned to one of two treatment conditions - 1. six months of weekly CPP intervention sessions OR 2. control condition in which mothers and their children will be referred for usual treatment in the community. Random assignment will be done based on a pre-determined schedule (a random number generator will be used to create a schedule for patient treatment assignment). Following randomization mother-child patient dyads will complete the following assessments: Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). All assessments will be conducted by a licensed clinician in conjunction with a research assistant.

Mothers (30 in each group) will be recruited through the Women's Program and pediatric practices affiliated with Columbia University Medical Center, including the Columbia Center of the New York Presbyterian Hospital, as well as its satellite center, the Allen Pavilion, and the Children's Hospital of New York. Approximately 90 women will need to screened to recruit 60 women for the study.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18-40 years
* Child age 3-5 years
* Maternal Beck Depression Inventory-II score 14-30
* Maternal report of at least two of ten child emotional/behavioral problems (excessive shyness, fussiness, sleep pattern problems, irritability, frequent inappropriate behavior) during phone screen administration of an adapted version of the Child Behavior Checklist.

Exclusion Criteria:

* Maternal lack of fluency in English as assessed through phone screening
* Maternal self-report of suicidality as assessed through Beck Depression Inventory-II
* Maternal self-report of Psychotic/Bipolar/Thought disorder
* Maternal self-report of substance abuse problems in the past 6 months
* Maternal report of child's lack of fluency in English
* Maternal report of child's developmental disorders / mental retardations / significant speech and language delays

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Symptoms of Depression (Beck Depression Inventory) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in maternal depression (Beck Depression Inventory) will assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). Assessments will be conducted by a licensed clinical psychologist in conjunction with a research assistant. Control variables i.e. daily stressors (Daily Hassles and Uplifts Scale), and social support (Social Support Questionnaire) will be assessed each time.
Change in Children's Emotional/Behavioral Functioning (Child Behavior Checklist) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in children's emotional and behavioral functioning (mother and a co-informant identified by the mother as someone who observes the child frequently will be asked to complete the Child Behavior Checklist) at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).

SECONDARY OUTCOMES:
Change in Children's Social Processes (NEuroPSYchological Assessment (NEPSY - II), Affect Recognition and Theory of Mind subtests) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in children's social processes (child performance on NEuroPSYchological Assessment (NEPSY - II), Affect Recognition and Theory of Mind subtests) will be assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).
Change in Maternal Parenting-Related Cognitions (Working Model of the Child Interview and Parenting Sense of Competence Scale) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in maternal parenting-related cognitions (Parenting Sense of Competence Scale) will be assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1), and via the Working Model of the Child Interview (WMCI) at Time 1 (pre-treatment) assessment, and Time 3 (after 24 sessions or an average of six months).
Change in Maternal Emotional Availability (free play coding using Emotional Availability scales) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in maternal emotional availability (free play coding using Emotional Availability scales will be assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). Mother and children will be asked to play together on a mat on the floor. Toys will be provided. Free play will be videotaped recorded for 15-20 minutes and later coded using the Emotional Availability (EA) scales. Two or more trained coders will code these play sessions.
Change in Children's Levels of Basal Cortisol (in Saliva) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Investigators will collect saliva samples from child (two saliva samples thirty minutes apart at each assessment) at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). Following each saliva collection, the swab will be placed into a salivette tube and frozen at -20°C or -80°C (per manufacturers instructions) until analysis. Once an adequate number of samples have been collected for analysis (to be determined by CRC), analysis will be run for levels of cortisol.
Change in Children's Levels of Immune Marker (C-Reactive Protein and Secretory Immunoglobulin A in Saliva) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  At the Time 1 interview on Day 1, and the second interview [Time 2, after 12 sessions or an average of three months], third interview [Time 3, after 24 sessions or an average of six months], and fourth interview [Time 4, six months after the completion of 24 treatment sessions or an average of one year after Time 1], the investigators will collect salivary samples from both mother and child. The investigators will collect two saliva samples from each child, thirty minutes apart during the assessment. Following each saliva collection, the swab will be placed into a salivette tube and frozen at -20°C or -80°C (per manufacturers instructions) until analysis.Once an adequate number of samples have been collected for analysis (to be determined by CRC), analysis will be run for levels of C-Reactive protein and Secretory Immunoglobulin A.
Change in Mothers' Levels of Basal Cortisol (in Saliva) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Investigators will collect saliva samples from mother (two saliva samples thirty minutes apart at each assessment) at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). Following each saliva collection, the swab will be placed into a salivette tube and frozen at -20°C or -80°C (per manufacturers instructions) until analysis. Once an adequate number of samples have been collected for analysis (to be determined by CRC), analysis will be run for levels of cortisol.
Change in Mothers' Levels of Immune Marker (C-Reactive Protein and Secretory Immunoglobulin A in Saliva) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Investigators will collect saliva samples from mother (two saliva samples thirty minutes apart at each assessment) at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1). Following each saliva collection, the swab will be placed into a salivette tube and frozen at -20°C or -80°C (per manufacturers instructions) until analysis. Once an adequate number of samples have been collected for analysis (to be determined by CRC), analysis will be run for levels of C-Reactive Protein and Secretory Immunoglobulin A.
Change in Maternal Global Symptoms of Distress (Symptom Checklist-90-R) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in maternal global symptoms of distress (Symptom Checklist-90-R) will assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).
Change in Maternal Post-Traumatic Stress Symptoms (Post-traumatic Diagnostic Scale) | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in maternal post-traumatic stress symptoms (Post-traumatic Diagnostic Scale) will assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).
Change in Child Mood and Post-Traumatic Stress Symptoms | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in children's mood and post-traumatic stress symptoms (child performance on Diagnostic Infant and Preschool Assessment (DIPA)) will be assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).
Change in Child's Executive Function | 1 year (six months after 24 session treatment or average of one year after pre-treatment assessment)
  Change in children's executive function (child performance on Behavior Rating Inventory of Executive Function will be assessed at Time 1 (pre-treatment) assessment, Time 2 (after 12 sessions or an average of three months), Time 3 (after 24 sessions or an average of six months), and Time 4 (six months after 24 treatment sessions or an average of one year after Time 1).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — New York State Psychiatric Institute, Columbia University Medical Center; Andrew Gerber, MD, Study Director — New York State Psychiatric Institute; Archana Basu, PhD, Study Director — Columbia University; Elizabeth Werner, PhD, Study Director — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Carpenter LL, Gawuga CE, Tyrka AR, Lee JK, Anderson GM, Price LH. Association between plasma IL-6 response to acute stress and early-life adversity in healthy adults. Neuropsychopharmacology. 2010 Dec;35(13):2617-23. doi: 10.1038/npp.2010.159. Epub 2010 Sep 29. PMID 20881945
- [Background] Chandra RK. Nutrition and the immune system from birth to old age. Eur J Clin Nutr. 2002 Aug;56 Suppl 3:S73-6. doi: 10.1038/sj.ejcn.1601492. PMID 12142969
- [Background] Chen E, Miller GE, Kobor MS, Cole SW. Maternal warmth buffers the effects of low early-life socioeconomic status on pro-inflammatory signaling in adulthood. Mol Psychiatry. 2011 Jul;16(7):729-37. doi: 10.1038/mp.2010.53. Epub 2010 May 18. PMID 20479762
- [Background] Coe CL, Laudenslager ML. Psychosocial influences on immunity, including effects on immune maturation and senescence. Brain Behav Immun. 2007 Nov;21(8):1000-8. doi: 10.1016/j.bbi.2007.06.015. Epub 2007 Aug 15. PMID 17706917
- [Background] Coe CL, Lubach GR. Critical periods of special health relevance for psychoneuroimmunology. Brain Behav Immun. 2003 Feb;17(1):3-12. doi: 10.1016/s0889-1591(02)00099-5. PMID 12615044
- [Background] Cole SW. Social regulation of leukocyte homeostasis: the role of glucocorticoid sensitivity. Brain Behav Immun. 2008 Oct;22(7):1049-1055. doi: 10.1016/j.bbi.2008.02.006. Epub 2008 Apr 3. PMID 18394861
- [Background] Danese A, Pariante CM, Caspi A, Taylor A, Poulton R. Childhood maltreatment predicts adult inflammation in a life-course study. Proc Natl Acad Sci U S A. 2007 Jan 23;104(4):1319-24. doi: 10.1073/pnas.0610362104. Epub 2007 Jan 17. PMID 17229839
- [Background] de Heredia FP, Gomez-Martinez S, Marcos A. Obesity, inflammation and the immune system. Proc Nutr Soc. 2012 May;71(2):332-8. doi: 10.1017/S0029665112000092. Epub 2012 Mar 20. PMID 22429824
- [Background] DeVries AC, Craft TK, Glasper ER, Neigh GN, Alexander JK. 2006 Curt P. Richter award winner: Social influences on stress responses and health. Psychoneuroendocrinology. 2007 Jul;32(6):587-603. doi: 10.1016/j.psyneuen.2007.04.007. Epub 2007 Jun 21. PMID 17590276
- [Background] Feder A, Alonso A, Tang M, Liriano W, Warner V, Pilowsky D, Barranco E, Wang Y, Verdeli H, Wickramaratne P, Weissman MM. Children of low-income depressed mothers: psychiatric disorders and social adjustment. Depress Anxiety. 2009;26(6):513-20. doi: 10.1002/da.20522. PMID 19016460
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Gouin JP, Glaser R, Malarkey WB, Beversdorf D, Kiecolt-Glaser JK. Childhood abuse and inflammatory responses to daily stressors. Ann Behav Med. 2012 Oct;44(2):287-92. doi: 10.1007/s12160-012-9386-1. PMID 22714139
- [Background] Irwin MR. Human psychoneuroimmunology: 20 years of discovery. Brain Behav Immun. 2008 Feb;22(2):129-39. doi: 10.1016/j.bbi.2007.07.013. Epub 2007 Oct 29. PMID 17911004
- [Background] Kurstjens S, Wolke D. Effects of maternal depression on cognitive development of children over the first 7 years of life. J Child Psychol Psychiatry. 2001 Jul;42(5):623-36. PMID 11464967
- [Background] Lieberman AF, Van Horn P, Ippen CG. Toward evidence-based treatment: child-parent psychotherapy with preschoolers exposed to marital violence. J Am Acad Child Adolesc Psychiatry. 2005 Dec;44(12):1241-8. doi: 10.1097/01.chi.0000181047.59702.58. PMID 16292115
- [Background] Lieberman AF, Ghosh Ippen C, VAN Horn P. Child-parent psychotherapy: 6-month follow-up of a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2006 Aug;45(8):913-918. doi: 10.1097/01.chi.0000222784.03735.92. PMID 16865033
- [Background] Murray L. The impact of postnatal depression on infant development. J Child Psychol Psychiatry. 1992 Mar;33(3):543-61. doi: 10.1111/j.1469-7610.1992.tb00890.x. PMID 1577898
- [Background] McDade TW. Early environments and the ecology of inflammation. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17281-8. doi: 10.1073/pnas.1202244109. Epub 2012 Oct 8. PMID 23045646
- [Background] Pace TW, Wingenfeld K, Schmidt I, Meinlschmidt G, Hellhammer DH, Heim CM. Increased peripheral NF-kappaB pathway activity in women with childhood abuse-related posttraumatic stress disorder. Brain Behav Immun. 2012 Jan;26(1):13-7. doi: 10.1016/j.bbi.2011.07.232. Epub 2011 Jul 27. PMID 21801830
- [Background] Schechter DS, Coots T, Zeanah CH, Davies M, Coates SW, Trabka KA, Marshall RD, Liebowitz MR, Myers MM. Maternal mental representations of the child in an inner-city clinical sample: violence-related posttraumatic stress and reflective functioning. Attach Hum Dev. 2005 Sep;7(3):313-31. doi: 10.1080/14616730500246011. PMID 16210242
- [Background] Schechter DS, Coates SW, Kaminer T, Coots T, Zeanah CH Jr, Davies M, Schonfeld IS, Marshall RD, Liebowitz MR, Trabka KA, McCaw JE, Myers MM. Distorted maternal mental representations and atypical behavior in a clinical sample of violence-exposed mothers and their toddlers. J Trauma Dissociation. 2008;9(2):123-47. doi: 10.1080/15299730802045666. PMID 18985165
- [Background] Scheeringa MS, Haslett N. The reliability and criterion validity of the Diagnostic Infant and Preschool Assessment: a new diagnostic instrument for young children. Child Psychiatry Hum Dev. 2010 Jun;41(3):299-312. doi: 10.1007/s10578-009-0169-2. PMID 20052532
- [Background] Shanahan L, Copeland WE, Worthman CM, Angold A, Costello EJ. Children with both asthma and depression are at risk for heightened inflammation. J Pediatr. 2013 Nov;163(5):1443-7. doi: 10.1016/j.jpeds.2013.06.046. Epub 2013 Aug 3. PMID 23919906
- [Background] Shonkoff JP. From neurons to neighborhoods: old and new challenges for developmental and behavioral pediatrics. J Dev Behav Pediatr. 2003 Feb;24(1):70-6. doi: 10.1097/00004703-200302000-00014. PMID 12584488
- [Background] Sohr-Preston SL, Scaramella LV. Implications of timing of maternal depressive symptoms for early cognitive and language development. Clin Child Fam Psychol Rev. 2006 Mar;9(1):65-83. doi: 10.1007/s10567-006-0004-2. PMID 16817009
- [Background] Toth SL, Rogosch FA, Manly JT, Cicchetti D. The efficacy of toddler-parent psychotherapy to reorganize attachment in the young offspring of mothers with major depressive disorder: a randomized preventive trial. J Consult Clin Psychol. 2006 Dec;74(6):1006-16. doi: 10.1037/0022-006X.74.6.1006. PMID 17154731
- [Background] Weissman MM, Pilowsky DJ, Wickramaratne PJ, Talati A, Wisniewski SR, Fava M, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Trivedi MH, Rush AJ; STAR*D-Child Team. Remissions in maternal depression and child psychopathology: a STAR*D-child report. JAMA. 2006 Mar 22;295(12):1389-98. doi: 10.1001/jama.295.12.1389. PMID 16551710